CLINICAL TRIAL: NCT01875484
Title: Impact of Circulating miR-126 on Left Ventricular Remodeling and Clinical Outcomes in Patients Undergoing Primary Percutaneous Coronary Intervention. The PMIR-miR-126 Study.
Brief Title: Circulating miR-126 as a Novel Biomarker for Post Myocardial Infarction Remodeling
Acronym: PMIR-miR-126
Status: Completed | Type: Observational
Sponsor: Qilu Hospital of Shandong University (Other)
Collaborators: Qianfoshan Hospital (Other); Jinan Central Hospital (Other); Shandong Provincial Hospital (Other Government); The Second Hospital of Shandong University (Other); Ruijin Hospital (Other); Qingdao University (Other); Shandong Provincial Medical Imaging Institute of Shandong University (Unknown); The First Affiliated Hospital of Zhengzhou University (Other); Heze Municipal Hospital (Other); Jining Hospital of Traditional Chinese Medicine (Other); Qihe People's Hospital (Unknown); Central Hospital of Zibo (Other); Weihai Municipal Hospital (Other); Beijing Friendship Hospital (Other); Binzhou Medical University (Other); Beijing Hospital (Other Government)
Responsible Party: Principal Investigator, Pan-Pan Hao, MD, PhD, Qilu Hospital of Shandong University
Other Study IDs: 2012CB518603
Record Dates: First submitted 2013-05-07; First posted 2013-06-11 (Estimated); Last update posted 2015-07-30 (Estimated); Status verified 2015-07

CONDITIONS: Myocardial Infarction; Left Ventricular Remodeling; miR-126
Keywords: miR-126; Left Ventricular Remodeling; Myocardial Infarction; primary percutaneous coronary intervention; left ventricular end diastolic volume; left ventricular ejection fraction; major adverse cardiovascular events
MeSH Terms: conditions — Myocardial Infarction; Ventricular Remodeling

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood Samples: serum, plasma, RNA, DNA, microRNAs, CD34+ cells
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- High miR-126 group
- Moderate miR-126 group
- Low miR-126 group

SUMMARY:
Purpose: The purpose of this study is to evaluate the impact of circulating miR-126 on left ventricular remodeling and clinical outcomes in patients undergoing primary percutaneous coronary intervention for ST-segment elevation myocardial infarction.

ELIGIBILITY:
Inclusion Criteria:

* Admitted for primary PCI for STEMI involving the LAD within 12 hours of onset of symptoms. STEMI will be defined as typical ECG changes (ST segment elevation ≥2mm in 2 or more precordial leads) associated with acute chest pain or an elevation of cardiac enzymes;
* Age ≥18 years;
* Informed consent from patient or next of kin.

Exclusion Criteria:

* Nonischaemic Cardiomyopathy;
* Cardiac surgery planed in the 6 months;
* Mechanical complication of STEMI (ventricular septal rupture, free wall rupture, acute severe mitral regurgitation);
* Renal or hepatic failure;
* Malignancy, HIV, or central nervous system disorder;
* Cardiopulmonary resuscitation >15 min and compromised level of consciousness;
* Cardiogenic shock;
* Current participation in any research study involving investigational drugs or devices;
* No written consensus;
* Previous myocardial infarction.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients undergoing primary PCI for STEMI
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Actual)
Dates: Start 2012-02; Primary Completion 2015-06 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Change in LVEDV from baseline by 3D-echocardiogram | 6 months
  The primary outcome of this study will be the change from baseline in left ventricular end diastolic volume (LVEDV) at 6 months post-PCI by 3D-echocardiogram.

SECONDARY OUTCOMES:
Major adverse cardiovascular events (MACE) | 6 months
  Cardiovascular death, myocardial infarction, target vessel revascularization,recurrent ischaemia, heart failure
All cause mortality | 6 months
Stent thrombosis | 6 months
Change in LVESV from baseline | 6 months
  Change from baseline in left ventricular end systolic volume (LVESV), ejection fraction (LVEF) and mass at 6 months post-PCI by 3D-echocardiogram
NT-proBNP levels | at 1 and 180 days post-PCI
Incidence of complete ST-segment resolution | 3 hours after PCI
Peak troponin T level | 24 hours after PCI

CONTACTS AND LOCATIONS:
Locations (17):
- China (17):
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Affiliated Hospital of Binzhou Medical Universty, Binzhou, Shandong
  - Heze Municipal Hospital, Heze, Shandong
  - Qianfoshan Hospital, Shandong University, Jinan, Shandong
  - Qilu Hospital, Shandong University, Jinan, Shandong
  - Jinan Central Hospital, Shandong University, Jinan, Shandong
  - Shandong Provincial Hospital, Shandong University, Jinan, Shandong
  - Shandong Provincial Medical Imaging Institute, Shandong University, Jinan, Shandong
  - The Second Hospital of Shandong University, Jinan, Shandong
  - Jining Hospital of Traditional Chinese Medicine, Jining, Shandong
  - Qihe People's Hospital, Qihe, Shandong
  - Affiliated Hospital of Qingdao University Medical College, Qingdao, Shandong
  - Weihai Municipal Hospital, Weihai, Shandong
  - Central Hospital of Zibo, Zibo, Shandong
  - Ruijin Hospital, School of Medicine, Shanghai Jiao Tong University, Shanghai, Shanghai Municipality
  - Beijing Friendship Hospital Affiliated to Capital Medical University, Beijing
  - Beijing Hospital, Beijing